CLINICAL TRIAL: NCT00023413
Title: TBTC Study 23C: Intensive Pharmacokinetic Study of Intermittent Rifabutin and Isoniazid With Daily Efavirenz in Combination With Two Nucleoside Analogs for Treatment of HIV and Tuberculosis Co-infections
Brief Title: TBTC Study 23C: Pharmacokinetics of Intermittent Rifabutin and Isoniazid With Daily Efavirenz
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-2588; 23C
Record Dates: First submitted 2001-09-06; First posted 2001-09-10 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: HIV Infections; Tuberculosis
Keywords: tuberculosis; TB
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Rifabutin; efavirenz

INTERVENTIONS:
Drug: Rifabutin
Drug: Efavirenz

SUMMARY:
The aim of this trial is to study the efavirenz-rifabutin interaction. Thus, this trial will enroll patients with HIV and tuberculosis co-infections who are receiving a rifabutin-based regimen and who plan to begin an antiretroviral regimen containing efavirenz dosed at 600 mg daily. Enrollment in TB Trials Consortium Study 23 is not a requirement for participation in this study.

Primary Objective:

To compare the pharmacokinetics of rifabutin at 600 mg twice a week in combination with efavirenz 600 mg daily to the pharmacokinetics of rifabutin 300 mg twice a week without efavirenz.

ELIGIBILITY:
* Patients with HIV and tuberculosis co-infections who are receiving a rifabutin-based regimen and who plan to begin an antiretroviral regimen containing efavirenz dosed at 600 mg daily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 1999-11; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Compare PK of rifabutin 600mg twice weekly with efavirenz 600mg daily to PK of rifabutin 300mg twice weekly without efavirenz

SECONDARY OUTCOMES:
*Describe PK of rifabutin 600mg twice weekly in combination with efavirenz 600mg daily with 2 NRTI's
*Describe PK of efavirenz in this regimen
*Assess safety of concomitant rifabutin and efavirenz in HIV-TB

CONTACTS AND LOCATIONS:
Overall Officials: Marc Weiner, MD, Principal Investigator — San Antonio VAMC, San Antonio TX
Locations (23):
- United States (20):
  - Central Arkansas Veterans Health System, Little Rock, Arkansas
  - LA County/USC Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Denver Department of Public Health and Hospitals, Denver, Colorado
  - Washington, D.C. VAMC, Washington D.C., District of Columbia
  - Chicago VA Medical Center (Lakeside), Chicago, Illinois
  - Hines VA Medical Center, Hines, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - New Jersey Medical School, Newark, New Jersey
  - New York University School of Medicine, New York, New York
  - Columbia University/Presbyterian Medical Center, New York, New York
  - Harlem Hospital Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Nashville VA Medical Center, Nashville, Tennessee
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Thomas Street Clinic, Houston, Texas
  - Audi L. Murphy VA Hospital, San Antonio, Texas
  - Seattle King County Health Department, Seattle, Washington
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Montreal Chest Institute McGill University, Montreal, Quebec

REFERENCES:
- See also: (Click here for more information about the Tuberculosis Trials Consortium(TBTC) — http://www.cdc.gov/nchstp/tb/tbtc/